CLINICAL TRIAL: NCT06397443
Title: Pronti A Salpare: Studio di fattibilità Sull'Impatto Della Vela Come Ergoterapia in Pazienti Con Malattie Rare Scheletriche - Ready to Sail: Evaluating Sailing's Feasibility as Ergotherapy for Rare Skeletal Diseases
Brief Title: Ready to Sail: Evaluating Sailing's Feasibility as Ergotherapy
Acronym: PaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Luca Sangiorgi, Director of the Rare Skeletal Disorders Department, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 115/2024/Sper/IOR
Record Dates: First submitted 2024-04-11; First posted 2024-05-02 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Multiple Osteochondroma; Ollier Disease; Osteogenesis Imperfecta
Keywords: Rare Diseases; QoL; Movement confidence; Mental health; Social interaction; Sailing
MeSH Terms: conditions — Exostoses, Multiple Hereditary; Enchondromatosis; Osteogenesis Imperfecta; Rare Diseases; Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with rare skeletal disorders (Experimental): 5-day sailing activity
  Interventions: Other: 5-day sailing activity

INTERVENTIONS:
Other: 5-day sailing activity — * Sailing activity (4 h/die)
  * Stretching exercises pre and post-sailing activity
  * Post-activity debriefing

SUMMARY:
Background Individuals with rare skeletal disorders frequently experience psychological distress, social isolation, unmet needs, and significant challenges due to limited treatment options. Adventure Therapy, employing exposure to natural environments, has shown promise in improving self-esteem, autonomy, and social skills in chronic illness and disability populations. This pilot study explores the feasibility and preliminary efficacy of a sailing-based intervention for enhancing physical, social, and psychological well-being in this specific population.

Outcome Measures The primary outcome is to investigates the feasibility of sailing to improve well-being and quality of life in patients living with rare skeletal disorders.

Furthermore, the investigators hypothesize that participation in a sailing program led by occupational therapists will lead to improvements in:

* Movement confidence: assessing whether sailing enhances participants' ability to move and perform daily activities.
* Mental health: evaluating if sailing reduces anxiety and fear and promotes self-esteem.
* Social interaction: exploring if sailing fosters social connection and reduces feelings of isolation.

Methods The study will use a prospective, single-arm, longitudinal design. Eight participants with rare skeletal disorders will be enrolled in a 5-day sailing-based occupational therapy intervention. Comprehensive pre- and post-intervention assessments will measure psychosocial factors, quality of life, functional mobility, kinesiophobia, and body segment movement using questionnaires and functional scales.

DETAILED DESCRIPTION:
Rare skeletal diseases represent a significant global health burden, affecting millions of people worldwide. These chronic, debilitating conditions necessitate the development of optimized clinical pathways and comprehensive support systems.

Adventure therapy (AT) has emerged as a promising intervention for individuals with chronic conditions, demonstrating improvements in self-esteem, autonomy, and social skills. Sailing, a form of AT, offers opportunities for physical activity, social inclusion, and emotional well-being in individuals with disabilities.

This study aims to assess the feasibility of using sailing as an occupational therapy intervention for patients with rare skeletal diseases. We hypothesize that sailing can enhance physical, cognitive, and social functioning in this patient population.

A pilot program of sailing lessons for patients with rare skeletal diseases will be conducted. Participants will undergo assessments of physical, cognitive, and social skills before and after the intervention.

This study will be the first to explore the use of sailing-based AT for this patient population. The findings will inform the development of larger-scale studies and contribute to the optimization of rehabilitation programs for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of any gender
* Diagnosis of a rare skeletal disease, confirmed clinically and/or molecularly
* Age 12 years or older
* No history of surgery within six months prior to study enrollment.

Exclusion Criteria:

* Individuals undergoing diagnostic evaluation for a rare skeletal disease
* Participants younger than 12 years of age.
* Individuals who underwent surgery within the preceding 6 months.
* Participants with fractures or musculoskeletal injuries sustained within the past year.
* Individuals who were unable to provide written informed consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MD, PhD, Principal Investigator — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cornaglia Ferraris P. [Adventure therapy: principles, practice, perspectives.]. Recenti Prog Med. 2018 Oct;109(10):487-493. doi: 10.1701/3010.30086. Italian. PMID 30394410
- [Background] MacLachlan M. Sailing as an Intervention. In: MacLachlan M, editor. Maritime Psychology: Research in Organizational & Health Behavior at Sea. Cham: Springer International Publishing; 2017. https://doi.org/10.1007/978-3-319-45430-6_10
- [Background] Thompson T, Lamont-Robinson C, Williams V. At sea with disability! Transformative learning in medical undergraduates voyaging with disabled sailors. Med Educ. 2016 Aug;50(8):866-79. doi: 10.1111/medu.13087. PMID 27402046
- [Background] Recio AC, Becker D, Morgan M, Saunders NR, Schramm LP, McDonald JW 3rd. Use of a virtual reality physical ride-on sailing simulator as a rehabilitation tool for recreational sports and community reintegration: a pilot study. Am J Phys Med Rehabil. 2013 Dec;92(12):1104-9. doi: 10.1097/PHM.0000000000000012. PMID 24252935
- [Background] Tracey D, Gray T, Truong S, Ward K. Combining Acceptance and Commitment Therapy With Adventure Therapy to Promote Psychological Wellbeing for Children At-Risk. Front Psychol. 2018 Aug 27;9:1565. doi: 10.3389/fpsyg.2018.01565. eCollection 2018. PMID 30210398
- [Background] Capurso, M.; Borsci, S. Effects of a Tall Ship Sail Training Experience on Adolescents' Self-Concept. International Journal of Educational Research 2013, 58, 15-24. https://doi.org/10.1016/j.ijer.2013.01.004.
- [Background] Gill E, Goldenberg M, Starnes H, Phelan S. Outdoor adventure therapy to increase physical activity in young adult cancer survivors. J Psychosoc Oncol. 2016 May-Jun;34(3):184-99. doi: 10.1080/07347332.2016.1157718. Epub 2016 Mar 3. PMID 26939742
- [Background] Zebrack B, Kwak M, Sundstrom L. First Descents, an adventure program for young adults with cancer: who benefits? Support Care Cancer. 2017 Dec;25(12):3665-3673. doi: 10.1007/s00520-017-3792-7. Epub 2017 Jun 27. PMID 28656467
- [Background] Aprile I, Iacovelli C, Iuvone L, Imbimbo I, Cruciani A, Pecchioli C, Manozzi FM, Padua L. Use of a Virtual-Technological Sailing Program to Prepare Children With Disabilities for a Real Sailing Course: Effects on Balance and Quality of Life. J Child Neurol. 2016 Jul;31(8):1074-80. doi: 10.1177/0883073816638756. Epub 2016 Mar 28. PMID 27021144
- [Derived] Boarini M, Banchelli F, Fittipaldi S, Scognamiglio D, Farella GM, Platano D, Rogati G, Di Sipio E, Villa G, Berti L, Leardini A, Sartini S, Scopinaro A, Sangiorgi L. Feasibility and safety of sailing based rehabilitation for rare skeletal disorders using wearable sensors and patient reported outcomes. Sci Rep. 2025 Oct 23;15(1):37153. doi: 10.1038/s41598-025-22231-8. PMID 41131085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was enrolled on May 16, 2024, and the last participant was also enrolled on May 16, 2024.
Pre-assignment Details: Of 10 eligibility participants, 8 met inclusion criteria and were included in the study.
Groups:
- Patients With Rare Skeletal Disorders: 5-day sailing activity
  5-day sailing activity: - Sailing activity (4 h/die)
  * Stretching exercises pre and post-sailing activity
  * Post-activity debriefing
Period: Overall Study
Arm/Group | Patients With Rare Skeletal Disorders
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 14 [12 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 8
Region of Enrollment [Number; unit: participants]
  Italy | 8

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life
Description: EuroQol 5-Dimension (EQ-5D) instrument offers valuable information about patient-reported health status. The questionnaire consists of two sections-descriptive system and visual analog scale (VAS)-and yields two scores: Index Value (IV), and overall health status (VAS).
  In the descriptive system section, patients report their level of problems in five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-and rate their health on a 5-level options for adults, and 3-level for adolescents and children. Based on the pattern of their responses, patients generate a health profile ranging from best health (11111 = highest level) to worst health (55555 = lowest level). Each health profile is transformed into an IV, that varies from 0 (absence of life/death) to 1 (perfect health).
  The VAS measures the patients' overall health status, with a score ranging from 0 ("The worst health you can imagine") to 100 ("The best health you can imagine").
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  EQ-5D Index Value | 0.91 [0.65 to 1]
  EQ-5D VAS | 84 [50 to 99]

2. Primary Outcome: Health-related Quality of Life
Description: as for outcome 1
Time Frame: T1: up to 2 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  EQ-5D Index Value | 0.91 [0.75 to 1]
  EQ-5D VAS | 90.50 [45 to 100]

3. Primary Outcome: Health-related Quality of Life
Description: as for outcome 1
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  EQ-5D Index Value | 0.90 [0.75 to 1]
  EQ-5D VAS | 93.50 [70 to 100]

4. Primary Outcome: Health-related Quality of Life
Description: as for outcome 1
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  EQ-5D Index Value | 0.82 [0.72 to 0.95]
  EQ-5D VAS | 83.50 [50 to 99]

5. Secondary Outcome: Self-esteem
Description: Rosenberg Self-Esteem Scale: 10-item scales, ranging from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 22 [9 to 26]

6. Secondary Outcome: Self-esteem
Description: as for outcome 5
Time Frame: T1: up to 2 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 21 [11 to 23]

7. Secondary Outcome: Self-esteem
Description: as for outcome 5
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 22 [10 to 25]

8. Secondary Outcome: Self-esteem
Description: Rosenberg Self-Esteem Scale is a 10-item scale that assesses the self-esteem, ranging from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 21 [11 to 30]

9. Secondary Outcome: Motor Coordination
Description: Performance Oriented Mobility Assesment (Tinetti Balance Scale) is an administered 16-item task-oriented test that measures gait and balance abilities, primarily to assess fall risk. It uses a 3-point ordinal scale of 0, 1 and 2. Gait is scored over 12 and balance is scored over 16. The total score (Fall Risk) ranges from 0 to 28, with higher scores indicating better balance and gait performance (19 or below=High risk of falls; 20-23=Moderate risk of falls; 24-28=Low risk of falls).
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Gait | 16 [15 to 16]
  Balance | 12 [10 to 12]
  Fall Risk | 28 [25 to 28]

10. Secondary Outcome: Motor Coordination
Description: as for outcome 9
Time Frame: T1: up to 2 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Gait | 12 [11 to 12]
  Balance | 16 [15 to 16]
  Fall Risk | 28 [26 to 28]

11. Secondary Outcome: Motor Coordination
Description: as for outcome 9
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Gait | 12 [12 to 12]
  Balance | 16 [16 to 16]
  Fall Risk | 28 [28 to 28]

12. Secondary Outcome: Motor Coordination
Description: as for outcome 9
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Gait | 12 [10 to 12]
  Balance | 16 [15 to 16]
  Fall Risk | 28 [25 to 28]

13. Secondary Outcome: Balance
Description: Berg Balance Scale is a 14-item objective measure that assesses static balance and fall risk, item-level scores range from 0-4, determined by ability to perform the assessed activity. The total score ranges from 0 to 56, with higher scores indicating better balance. A score of less than 45 suggests an increased risk of falling.
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 56 [56 to 56]

14. Secondary Outcome: Balance
Description: as for outcome 13
Time Frame: T1: up to 2 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 56 [56 to 56]

15. Secondary Outcome: Balance
Description: as for outcome 13
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 56 [56 to 56]

16. Secondary Outcome: Balance
Description: as for outcome 13
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale | 56 [56 to 56]

17. Secondary Outcome: Kinesiophobia
Description: The Tampa Scale for Kinesiophobia (TSK) is a validated self-report questionnaire designed to assess the fear of movement or (re)injury in individuals experiencing pain or musculoskeletal disorders. The TSK consists of 13 items (Italian validated version), each rated on a 4-point Likert scale, ranging from 1 ("Strongly Disagree") to 4 ("Strongly Agree"). The scores are summed to yield a total score ranging from 13 to 52, with higher scores indicating greater levels of kinesiophobia.
  The TSK includes two subscales: 1.Activity Avoidance, with a score ranging from 6 to 24; 2.Harm Beliefs, with a score ranging from 7 to 28.
  Higher scores on both the Activity Avoidance and Harm Beliefs subscales indicate greater levels of kinesiophobia, reflecting increased fear of movement due to injury concerns (Activity Avoidance subscale) or harmful beliefs about physical activity (Harm Beliefs subscale).
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Activity Avoidance Scale | 10 [6 to 17]
  Harm Scale | 11 [8 to 18]
  Kinesiophobia | 21.50 [15 to 35]

18. Secondary Outcome: Kinesiophobia
Description: as for outcome 17
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Activity Avoidance Scale | 11 [7 to 16]
  Harm Scale | 12 [10 to 17]
  Kinesiophobia | 22.50 [19 to 30]

19. Secondary Outcome: Kinesiophobia
Description: as for outcome 17
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Activity Avoidance Scale | 10.50 [7 to 17]
  Harm Scale | 8 [5 to 11]
  Kinesiophobia | 18.50 [12 to 28]

20. Secondary Outcome: Well-being and Mental Health
Description: Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report questionnaire designed to assess psychological distress and monitor treatment response. It consists of 34 items evaluating emotional state and perceived well-being over the past week, rated on a 5-point Likert scale from 0 ("Not at all") to 4 ("Most or all of the time").
  The total score is calculated as the mean of all item scores and can be reported in two ways: 1.Raw score: The mean of all item scores (range: 0-4). 2.Standardized score: Obtained by multiplying the raw score by 10, yielding a scale from 0 to 40.
  The data presented in the results refer to the raw score.
  Score Interpretation:
  0.00-0.99: No clinical distress or minimal risk. 1.00-1.99: Mild distress, potentially significant. 2.00-2.99: Moderate distress, generally indicative of the need for intervention.
  3.00-4.00: Severe distress, highly indicative of the need for immediate clinical intervention.
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
units on a scale | 0.85 [0.10 to 2.70]

21. Secondary Outcome: Well-being and Mental Health
Description: as for outcome 20
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
units on a scale | 0.45 [0.10 to 1.60]

22. Secondary Outcome: Well-being and Mental Health
Description: as for outcome 20
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
units on a scale | 1.25 [0.60 to 2.30]

23. Secondary Outcome: Physical Functioning and Psychological Well-being
Description: Pediatric Outcomes Data Collection (PODCI) evaluates functional health status through an 83-item questionnaire, and uses domain-specific scales. Each scale generates a score ranging from 0 to 100, with higher scores indicating better functioning or less impairment.
Time Frame: T0: Baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Upper Extremity Scale | 95.83 [54.17 to 100]
  Transfer & Basic Mobility Scale | 92.80 [87.88 to 100]
  Sports and Physical Functioning Scale | 73.96 [58.33 to 100]
  Pain/Comfort Scale | 81.11 [46.11 to 100]
  Happiness Scale | 85 [55 to 100]
  Global Functioning Scale | 84.68 [69.65 to 100]

24. Secondary Outcome: Physical Functioning and Psychological Well-being
Description: as for outcome 23
Time Frame: T1: up to 2 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Upper Extremity Scale | 97.92 [66.67 to 100]
  Transfer & Basic Mobility Scale | 97.35 [87.88 to 100]
  Sports and Physical Functioning Scale | 81.53 [59.72 to 97.22]
  Pain/Comfort Scale | 71.39 [47.78 to 100]
  Happiness Scale | 82.50 [40 to 95]
  Global Functioning Scale | 86.71 [71.79 to 98.96]

25. Secondary Outcome: Physical Functioning and Psychological Well-being
Description: as for outcome 23
Time Frame: T2: up to 3 weeks
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Upper Extremity Scale | 97.92 [83.33 to 100]
  Transfer & Basic Mobility Scale | 97.35 [87.88 to 100]
  Sports and Physical Functioning Scale | 81.94 [48.48 to 100]
  Pain/Comfort Scale | 83.61 [49.44 to 100]
  Happiness Scale | 92.50 [40 to 100]
  Global Functioning Scale | 86.40 [79.91 to 100]

26. Secondary Outcome: Physical Functioning and Psychological Well-being
Description: as for outcome 23
Time Frame: T3: up to 3 months
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Patients With Rare Skeletal Disorders
Number analyzed (Participants) | 8
score on a scale
  Upper Extremity Scale | 97.92 [75 to 100]
  Transfer & Basic Mobility Scale | 96.97 [91.67 to 100]
  Sports and Physical Functioning Scale | 88.19 [51.39 to 97.50]
  Pain/Comfort Scale | 67.22 [38.33 to 93.33]
  Happiness Scale | 80 [55 to 100]
  Global Functioning Scale | 85.73 [77.10 to 97.50]

27. Other Pre Specified Outcome: Information on the Functioning and Disability of an Individual
Description: Functional Independence Measure (FIM) is a validated clinician-administered tool designed to assess functional independence in individuals with neurological or musculoskeletal conditions. It evaluates the level of assistance required for daily activities across six domains: self-care, sphincter control, mobility, locomotion, communication, and social cognition. The FIM consists of 18 items, each rated on a 7-point ordinal scale (1 = total assistance, 7 = complete independence), with total scores ranging from 18 to 126. Higher scores indicate greater functional independence.
Time Frame: T0
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Information on the Functioning and Disability of an Individual
Description: as for outcome 27
Time Frame: T3
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Kinesiophobia
Description: as for outcome 17
Time Frame: T1
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Well-being and Mental Health
Description: Clinical Outcomes in Routine Evaluation-Outcome Measure (CORE-OM) is a self-report measure of psychological distress designed to be administered during a course of treatment to determine treatment response. It compries 34 questions about how the participants have been feeling over the last week, using a 5-point Likert scale ranging from 0 ("Not at all") to 4 ("Most or all of the time"). The total score is calculated as the mean of all item scores (ranging from 0 to 4) and can be reported either as a raw score or standardized (e.g., multiplying the mean by 10 to obtain a score on a 0-40 scale).
  Score Interpretation:
  0-0.99: No clinical distress or minimal risk. 1.00-1.99: Mild distress, potentially significant. 2.00-2.99: Moderate distress, generally indicative of a need for intervention. 3.00-4.00: Severe distress, highly indicative of immediate clinical intervention.
Time Frame: T1
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Patients With Rare Skeletal Disorders
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT06397443/Prot_SAP_000.pdf